CLINICAL TRIAL: NCT00675844
Title: An Open-Label Treatment Protocol to Provide Continued Elvucitabine Treatment for 48 Weeks in Participants Who Have Completed 96 Weeks of Elvucitabine Therapy in Protocol ACH443-015 or 48 Weeks of Therapy in Protocol ACH443-018
Brief Title: An Open-Label Treatment Protocol to Provide Continued Elvucitabine Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: Achillion, a wholly owned subsidiary of Alexion (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACH443-904
Record Dates: First submitted 2008-05-08; First posted 2008-05-12 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: HIV Infections
Keywords: Extension study; HIV-1 infection; Treatment naive
MeSH Terms: conditions — HIV Infections | interventions — dexelvucitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Elvucitabine (Experimental): Participants currently receiving elvucitabine will continue elvucitabine as part of their antiretroviral therapy (ART) regimen for an additional 48 months.
  Interventions: Drug: Elvucitabine

INTERVENTIONS:
Drug: Elvucitabine — 10 milligrams (mg) elvucitabine daily as part of an ART regimen

SUMMARY:
Extension study for participants currently participating in Protocols ACH443-015 and ACH443-018.

DETAILED DESCRIPTION:
Human immunodeficiency virus (HIV)-1-infected, clinically stable, treatment-naïve adult participants who have completed 96 weeks of elvucitabine therapy and whose HIV ribonucleic acid (RNA) levels remain below 50 copies/milliliter (mL) at the 92-week assessment in Protocol ACH443-015 or participants who have completed 48 weeks of elvucitabine therapy and continue to maintain an HIV-1 RNA viral load below their baseline level upon entry into Protocol ACH443-018.

ELIGIBILITY:
Inclusion Criteria:

• Participants must have successfully completed 96 weeks of elvucitabine therapy in Protocol ACH443-015 or participants have completed 48 weeks of elvucitabine therapy in Protocol ACH443-014A-018 .

Exclusion Criteria:

* Participant has experienced virologic rebound as defined in Section 5.6.1.3 of Protocol ACH443-015.
* Participant has exceeded their Baseline HIV-1 RNA level by Week 44 as measured in Protocol ACH443-014A-018
* Participant is experiencing a drug-related Grade 3 or 4 rash or a drug-related Grade 3 or 4 laboratory toxicity other than Grade 3 or 4 cholesterol, triglyceride, creatinine kinase, or lactate dehydrogenase (LDH).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2008-05; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Determine Safety Profile Of Elvucitabine Measured By Incidence Of Study Discontinuations And Incidence, Severity, And Type Of Adverse Events And Clinically Significant Changes Or Abnormalities In Participant's Clinical Laboratory Results. | 48 months

SECONDARY OUTCOMES:
Determination Of The Continued Efficacy Of Elvucitabine As Measured By The Change In Helper T Cell (CD4) Count. | 48 months

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Clinical Trial Site, Orlando, Florida
  - Clinical Trial Site, Pensacola, Florida
  - Clinical Trial Site, Newark, New Jersey
  - Clinical Trial Site, Austin, Texas
  - Clinical Trial Site, Dallas, Texas